CLINICAL TRIAL: NCT03023306
Title: Effectiveness of Preemptive Versus Preventive Antiemetic Treatment in Patients Undergoing Laparoscopic Cholecystectomy. A Randomized Double Blind Trial.
Brief Title: Preemptive Versus Preventive Antiemetic Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Argyro Fassoulaki, Professor Emeritus, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB No 65/19-06-18
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preemptive group (Active Comparator): The preemptive group will receive the anti-emetic regimen i.v. (4 mg of ondansetron) 1h before the start of surgery. During surgery, 30 min before the end of operation, this group will receive i.v. 0.9% NaCl in equal volumes.The intervention consists of the different time points of antiemetic treatment, thus 1h before surgery vs intraopertively.
  Intervention: Antiemetic treatment 1h before surgery
  Interventions: Other: Antiemetics perioperatively
- intraoperative group (Other): The preventive group will receive i.v. 0.9% NaCl 1h before surgery and ondansetron 4 mg 30 min before the end of surgery at equal volumes.
  Intervention: Antiemetic treatment intraoperatively
  Interventions: Other: Antiemetics perioperatively

INTERVENTIONS:
Other: Antiemetics perioperatively — Preemptive group ondansetron 4 mg will be administered 1h before surgery Intraoperative group Ondansetron 4 mg will be administered intraoperatively

SUMMARY:
Patients aged between 20 and 70 years, ASA physical status I-III, and scheduled for laparoscopic cholecystectomy under general anaesthesia will be enrolled in the study.

Patients will be randomized to the preemptive group to receive an antiemetic regime 1h before the start of surgery or to the intraoperative group to receive the same antiemetic drugs in the same doses intraoperatively, 30 min before the end of surgery.

In the operating room standard monitoring and a standardized anesthetic technique will be implemented in all patients. Nausea, vomiting, retching and PONV (cumulative) will be recorded at PACU, at 4h, 8h and 24h postoperatively. Pain scores assessed by NRS (numerical rating scale) will be recorded at the same time points. Also, when patients received fluids and solid food by mouth will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III patients
* Surgical procedure: scheduled for laparoscopic cholecystectomy
* Type of anesthesia: general

Exclusion Criteria:

* Antihistamines the last three days
* Antiemetic drugs the last three days
* Hiatus hernia
* reflux
* Gastrointestinal disease
* Pregnancy
* BMI > 35
* parkinson
* known allergy to the drugs of the protocol
* epilepsy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
PONV (postoperative nausea vomiting combined) | 24 hours
  Incidence of combined nausea and vomiting postoperatively

SECONDARY OUTCOMES:
postoperative nausea frequency and intensity | 24 hours
  numerical rating scale of nausea intensity (0-10)
postoperative vomiting frequency | 24 hours
  number of vomits
postoperative pain | 24 hours
  numerical rating scale of pain intensity (0-10)
retching | 24 hours
  if retching exists
PONV (postoperative nausea vomiting combined) | 24 hours
  frequency and intensity of nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Aretaieio University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Odom-Forren J, Rayens MK, Gokun Y, Jalota L, Radke O, Hooper V, Wiggins AT, Apfel CC. The Relationship of Pain and Nausea in Postoperative Patients for 1 Week After Ambulatory Surgery. Clin J Pain. 2015 Oct;31(10):845-51. doi: 10.1097/AJP.0000000000000170. PMID 25370136
- [Background] Gan TJ, Diemunsch P, Habib AS, Kovac A, Kranke P, Meyer TA, Watcha M, Chung F, Angus S, Apfel CC, Bergese SD, Candiotti KA, Chan MT, Davis PJ, Hooper VD, Lagoo-Deenadayalan S, Myles P, Nezat G, Philip BK, Tramer MR; Society for Ambulatory Anesthesia. Consensus guidelines for the management of postoperative nausea and vomiting. Anesth Analg. 2014 Jan;118(1):85-113. doi: 10.1213/ANE.0000000000000002. PMID 24356162
- [Background] Apfel CC, Heidrich FM, Jukar-Rao S, Jalota L, Hornuss C, Whelan RP, Zhang K, Cakmakkaya OS. Evidence-based analysis of risk factors for postoperative nausea and vomiting. Br J Anaesth. 2012 Nov;109(5):742-53. doi: 10.1093/bja/aes276. Epub 2012 Oct 3. PMID 23035051
- [Background] Apfel CC, Meyer A, Orhan-Sungur M, Jalota L, Whelan RP, Jukar-Rao S. Supplemental intravenous crystalloids for the prevention of postoperative nausea and vomiting: quantitative review. Br J Anaesth. 2012 Jun;108(6):893-902. doi: 10.1093/bja/aes138. PMID 22593126
- [Background] Wallden J, Flodin J, Hultin M. Validation of a prediction model for post-discharge nausea and vomiting after general anaesthesia in a cohort of Swedish ambulatory surgery patients. Eur J Anaesthesiol. 2016 Oct;33(10):743-9. doi: 10.1097/EJA.0000000000000473. PMID 27270883
- [Derived] Theodosopoulou P, Staikou C, Fassoulaki A. Preoperative versus intraoperative antiemetic strategies in patients undergoing laparoscopic cholecystectomy: A randomised double-blind study. Eur J Anaesthesiol. 2023 Oct 1;40(10):769-776. doi: 10.1097/EJA.0000000000001888. Epub 2023 Jul 19. PMID 37466110